CLINICAL TRIAL: NCT04437823
Title: Efficacy of Intravenous Infusions of Stem Cells in the Treatment of COVID-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jinnah Hospital (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Prof. Sheikh Riazuddin, Distinguished National Professor, Jinnah Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JB&RSC-01
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Corona Virus Infection
Keywords: COVID-19; Stem Cells treatment
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Group 1 (15 subjects) Fifteen (15) subjects will be treated with three intravenous infusion (IV) of 5 x 10^5 (per Kg body weight) UCMSCs delivered via peripheral intravenous infusion on days 1, 3 and 5 besides the standard care (SOC).
  Group 2 (5 subjects) Five (5) subjects will be treated under SOC. From two subjects in group 1 will not be treated 24hrs apart. Patients will be randomized in a 1:3 ratio (SOC: UCMSC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : Treatment (Experimental): Fifteen (15) subjects will be treated with three intravenous infusion (IV) of 5 x 10^5 UCMSCs per Kg body weight delivered via peripheral intravenous infusion on days 1, 3 and 5 besides the standard care (SOC).
  Interventions: Biological: Intravenous Infusions of Stem Cells
- Group 2: standard care (No Intervention): Five (5) subjects will be treated under Standard of Care (SOC) .

INTERVENTIONS:
Biological: Intravenous Infusions of Stem Cells — Cultured stem cells will be injected at days 1, 3 and 5 intravenously. While patients will be monitored and evaluated for various hematological and organ functions at baseline (day 0) and days 1, 3, 5, 7, 14, 21 and 30
  Arms: Group 1 : Treatment

SUMMARY:
Stem cell therapy has emerged as a revolutionary treatment for diseases that were considered untreatable only a few years ago. Umbilical cord-derived mesenchymal stem cells (UCMSCs) have been shown to repair damaged liver, kidney, heart, pancreas, skin, cartilage, and cornea in animal models and several human trials. In addition to cellular replacement through regeneration, UCMSCs mediate through paracrine signaling pathways resulting in immune modulation. Clinical manifestations of coronavirus disease 2019 (COVID-19), are believed to arise from septic shock and cytokine storm that cause acute respiratory dysfunction and acute cardiac injury. There is presently no cure for the COVID-19 viral disease; however, multi-treatment strategies are being examined. During the past two months, four reports were published that suggest, mesenchymal stem cells (MSCs), owing to their powerful immunomodulatory ability, may prevent the cytokine storm and thus reduce the COVID-19 related morbidity. All studies reported that COVID-19 patients responded favorably to MSCs therapy. These reports, taken together with the previous successes of stem cell therapy in animal models, the investigators, a seven-institution consortium, propose to explore the efficacy of UCMSC treatment in COVID-19 patients at Jinnah hospital, Lahore. The investigators propose to administer UCMSCs in patients with acute pulmonary inflammation due to COVID-19 infection with moderate to severe symptoms. In the first cohort of 15 patients, UCMSCs will be administered with three intravenous infusions of 500,000 UCMSCs per Kg body weight each on days 1, 3, and 5. The second group of five patients serving as control will only receive standard treatment. During the 30-day post-infusion period, a battery of tests will be performed to evaluate the safety and efficacy of the UCMSCs treatment. In parallel, the investigators propose a comparative study to determine COVID-19 viral count by quantitative real-time PCR and through viral coat protein ELISA, developed in the investigator advisor lab (Dr. Tauseef Butt, Progenra Inc. Philadelphia, USA) with the ultimate objective to locally developing a rapid diagnostic assay.

DETAILED DESCRIPTION:
Isolation and characterization of human umbilical cord-derived mesenchymal stem cells (UCMSCs): Human umbilical cord tissues along with informed consent forms will be collected from hepatitis B, C, and COVID-19 virus-negative women with healthy pregnancies during the Cesarean Section surgery after completion of gestation period. The cord tissue will be transported in sterile 1x phosphate-buffered saline (PBS) containing 200 units/ml penicillin and 200 µg/ml streptomycin on ice. In the biosafety cabinet, the cord will be washed with 4-5 changes of sterile 1x PBS and placed in a Petri plate with 15 ml PBS. The cord will be gently scraped with a surgical blade to remove any dead cells. A 9 cm umbilical cord will be cut into three equal pieces and wash thoroughly to remove blood clots, umbilical cord arteries, and veins. Segments will be washed three times with PBS and minced. The minced pieces will be incubated in 17.5 ml of collagenase solution (201 U/ml collagenase type I in serum-free DMEM-HG) in a 50 ml conical tube for ~3.5 hours in an incubator at 5% CO2, 95% humidity at 37⁰C. After ~3.5 hours, the digested lysate will pass through a strainer and will be diluted three times with 1x PBS. Following centrifugation, the cells will be seeded into two 25 cm2 flasks and will be placed in an incubator at 5% CO2, 95% humidity at 37⁰C. The flasks will be fed with fresh media (DMEM-HG supplemented with 20% FBS and 1% antibiotic solution) every third day. At around day 18, cells will reach up to 85% confluency and will be transferred in two 75 cm2 flasks with media replaced at alternate days. UCMSCs at P3 will be characterized using different specific antibodies. Cells at P3 will be used for transplantation in patients. Fifteen (15) subjects will be treated with three intravenous infusions (IV) of 500,000 UCMSCs per Kg body weight delivered via peripheral intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Male or female subjects age >18 years at the time of signing the Informed Consent Form
* Must have a clinical diagnosis of COVID-19, with at least one of clinical symptoms (e.g., fever ≥38°C, fatigue, cough) and a positive result by the reverse-transcription polymerase chain reaction (RT-PCR) testing or equivalent
* Individuals with moderate to severe COVID-19 symptoms
* Adequate venous access
* For female patients only, willingness to use recommended birth control until 6 months post-treatment
* Must agree to comply with all study requirements and be willing to complete all study visits
* Need in-patient admission

Exclusion Criteria:

* A female who is pregnant, nursing, or of child-bearing potential while not practicing effective contraceptive methods. Female subjects must undergo a blood pregnancy test at screening and prior to infusion.
* Inability to perform any of the assessments required for endpoint analysis
* Have known allergies to penicillin or streptomycin
* Have a clinical history of malignancy within 3 years (i.e., subjects with prior malignancy must be disease-free for 3 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma, if recurrence occurs; - History of drug abuse (illegal "street" drugs except for marijuana, or prescription medications not being used appropriately for a pre-existing medical condition) or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months
* Be serum positive for HIV, hepatitis BsAg or Viremic hepatitis C.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy assessment of infusion associated adverse events | Day 01 to Day 30
  Number of participants with significant side effects in stem cell treated group
Chest Radiograph or Chest CT Scan | Day 01 to Day 30
  Assessment of Pneumonia improvement as a result of stem cell infusions

SECONDARY OUTCOMES:
COVID-19 Quantitative Real Time PCR | Day 01 to Day 30
  Quantitative real-time PCR analysis for the evaluation of negative corona virus test results following stem cell treatment
Sequential Organ Failure Assessment (SOFA) Score | Day 01 to Day 30
  Evaluation of organ function (Each organ system is assigned a value for 0 (normal) to 4 (highest degree of dysfunction))
Rate of mortality | Day 01 to Day 30
  Number of all mortalities within 30 days post first infusion
Clinical Respiratory Changes | Day 01 to Day 30
  Examination of improvement in the physiology of lungs after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Moazzam N Tarar, MBBS, FCPS, Principal Investigator — Jinnah Burn & Reconstructive Surgery Center, Lahore; Azra Mehmood, PhD, Principal Investigator — Centre of Excellence in Molecular Biology, Lahore
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The report will be published and available online.
Supporting Information: Study Protocol, CSR
Time Frame: At the end of completion of the study
Access Criteria: Available online

REFERENCES:
- [Background] Leng Z, Zhu R, Hou W, Feng Y, Yang Y, Han Q, Shan G, Meng F, Du D, Wang S, Fan J, Wang W, Deng L, Shi H, Li H, Hu Z, Zhang F, Gao J, Liu H, Li X, Zhao Y, Yin K, He X, Gao Z, Wang Y, Yang B, Jin R, Stambler I, Lim LW, Su H, Moskalev A, Cano A, Chakrabarti S, Min KJ, Ellison-Hughes G, Caruso C, Jin K, Zhao RC. Transplantation of ACE2- Mesenchymal Stem Cells Improves the Outcome of Patients with COVID-19 Pneumonia. Aging Dis. 2020 Mar 9;11(2):216-228. doi: 10.14336/AD.2020.0228. eCollection 2020 Apr. PMID 32257537
- [Background] Atluri S, Manchikanti L, Hirsch JA. Expanded Umbilical Cord Mesenchymal Stem Cells (UC-MSCs) as a Therapeutic Strategy in Managing Critically Ill COVID-19 Patients: The Case for Compassionate Use. Pain Physician. 2020 Mar;23(2):E71-E83. PMID 32214286
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119
- [Background] Riazuddin S et al.,. Book chapter: Stem cells for the repair of damaged skin and cartilage, in Book: Stem Cells - From Drug to Drug Discovery. Ed. by Haider, Khawaja Husnain; ISBN# 978-3-11-049376-4; March 2017
- [Background] Riazuddin S et al., Cell therapy for liver regeneration. In , (Eds.), Stem Cells - From Hype to Real Hope (pp. 130-145). Berlin, Boston: De Gruyter. https://doi.org/10.1515/9783110587043-007; Book DOI: https://doi.org/10.1515/9783110587043; Online ISBN: 9783110587043; © 2018 Walter de Gruyter GmbH, Berlin/Munich/Boston.